CLINICAL TRIAL: NCT00599326
Title: Pilot Trial of Deferasirox in the Treatment of Porphyria Cutanea Tarda
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Amit Pandya, Professor of Dermatology, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CICL670A US17; IRB File Number 062007-047
Record Dates: First submitted 2008-01-10; First posted 2008-01-23 (Estimated); Results first posted 2014-02-10 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2014-01

CONDITIONS: Porphyria Cutanea Tarda
Keywords: Exjade PCT Study; PCT Study; Porphyria Cutanea Tarda
MeSH Terms: conditions — Porphyria Cutanea Tarda | interventions — Deferasirox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: Deferasirox

INTERVENTIONS:
Drug: Deferasirox — 250 mg of deferasirox once daily for 6 months
  Other Names: Exjade

SUMMARY:
To determine the efficacy and tolerability of deferasirox in the treatment of Porphyria Cutanea Tarda.

Primary objective - the elimination of all blistering within 6 months of treatment.

Secondary objective - decrease in total body iron levels.

DETAILED DESCRIPTION:
Phlebotomy is the standard therapy for Porphyria Cutanea Tarda (PCT), but it can be inconvenient and cause anemia in some patients.

Deferasirox is a new class of tridentate iron chelators with high affinity and selectivity for iron. The medication is administered orally, which if effective for PCT would make it a more convenient and possibly more tolerable option for patients.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Porphyria Cutanea Tarda based on clinical exam and 24-hour urine porphyrin levels
* have Porphyria Cutanea Tarda for at least 3 months prior to enrollment with active blistering (3 blisters or erosions per month)
* women of childbearing potential must use an effective method of contraception during the study, however this cannot include hormonal contraception (oral contraceptives, hormone patches, Depo-Provera injections, NUVA Ring, etc.)
* treatment naive patients or patients unresponsive or intolerant of phlebotomy
* Ferritin level is greater than or equal to 25ng/mL

Exclusion Criteria:

* patients with serum creatinine above the upper limit of normal
* patients receiving phlebotomy who are controlled on this therapy
* pregnant or breast feeding females
* patients with liver transaminases more than 5 times the upper limit of normal
* patients with a history of hypersensitivity to deferasirox
* patients with a history of pre-existing renal condition, or receiving medication that depresses renal function
* patients on other chelators
* history of non-compliance to medical regimens.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Pandya, M.D., Principal Investigator — UT Southwestern Medical Center at Dallas - Department of Dermatology
Locations (1):
- UT Southwestern Medical Center at Dallas - Dermatology Clinical Trials, Dallas, Texas, United States

REFERENCES:
- [Derived] Pandya AG, Nezafati KA, Ashe-Randolph M, Yalamanchili R. Deferasirox for porphyria cutanea tarda: a pilot study. Arch Dermatol. 2012 Aug;148(8):898-901. doi: 10.1001/archdermatol.2012.807. PMID 22911183

RESULTS

PARTICIPANT FLOW:
Groups:
- Deferasirox: Deferasirox : 250 mg of deferasirox once daily for 6 months with an increase to 500 mg/d after 2 months if new blisters continued to develop.
Period: Overall Study
Arm/Group | Deferasirox
Started | 10
Completed | 8
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Noncompliant | 1

BASELINE CHARACTERISTICS:
Arm/Group | Deferasirox
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (5.907622195)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Showing Reduction or Elimination of Skin Blistering
Description: The present trial was undertaken to determine if oral deferasirox could be useful in the treatment of PCT. Monthly clinic visits with a physical examination was conducted to assess the skin for blisters.
Time Frame: Within 6 months of treatment.
Measure: Number; unit: participants
Arm/Group | Deferasirox
Number analyzed (Participants) | 8
participants
  Elimination | 0
  Reduction | 8

2. Secondary Outcome: Number of Participants Showing Decrease in Ferritin and Urinary Porphyrin Level
Description: Patients with PCT usually have normal or elevated serum iron and ferritin levels as well as increased iron absorption. Phlebotomy is conducted to analyzes the ferritin levels. Urine collection is performed and samples of the urine are analyzed for porphyrin levels.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Deferasirox
Number analyzed (Participants) | 8
participants
  Decrease in ferritin level | 8
  Decrease in urinary porphyrin level | 6

ADVERSE EVENTS:
Arm/Group | Deferasirox
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deferasirox (N=10)
Abdominal pain (Mild) (Gastrointestinal disorders) | 1 (1) — mild abdominal discomfort for 2 days in 1 patient, which resolved spontaneously.

LIMITATIONS AND CAVEATS:
10 patients were enrolled, of which 8 were compliant with therapy and had evaluable data. Of the 2 patients dropped from the study, one patient was lost to follow-up after 2 months and another was noncompliant with medication dosing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes